CLINICAL TRIAL: NCT04863196
Title: EFFECT OF LASER THERAPY ON MUCOSAL LESIONS OF GASTRIC STOMA OF CHILDREN AND ADOLESCENTS: RANDOMIZED CLINICAL TRIAL
Brief Title: LASER THERAPY IN GASTRIC STOMA INJURIES OF CHILDREN AND ADOLESCENTS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAAE30991020.0.0000.0068
Record Dates: First submitted 2021-02-26; First posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-02

CONDITIONS: Gastrostomy Complications
Keywords: Gastrostomy; Child; Adolescent; Laser therapy; Low-Level Light Therapy; Peristomal lesions; Nursing care

STUDY DESIGN:
Intervention Model Description: Randomized, open clinical trial to assess the healing time of a lesion present in the gastric stoma mucosa using laser therapy or protective barrier powder.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser therapy Treatment Group (Experimental): Treatment evaluation and follow-up will be done for 15 days. The application of the laser at first will be done three times a week.
  The application will be by points with continuous or selective technique, which will depend on each patient. The device is a pen type that will be by contact or without contact with the lesion, irradiation and the dose will be according to the calculation for each patient, using power in milliwatt and fluency, where the dose will vary according to area and patient, and may vary from 0.1 to 1J / cm² as calculated.
  The laser tip will be disinfected before each use with 70% alcohol and later coated with plastic film. Patients, companion and operator will wear specific eye protection glasses and all biosafety rules will be followed during therapy.
  Interventions: Other: Laser therapy Treatment Group
- Barrier Dust Treatment Group (Active Comparator): The evaluation and follow-up of the treatment will be done for 15 days. The principle application will be made three times a week using the protective barrier powder over the entire affected area, forming a protective barrier when adhering to the skin.
  For all patients, the injured area will be previously cleaned with 0.9% saline solution.
  Interventions: Other: Barrier Dust Treatment Group

INTERVENTIONS:
Other: Laser therapy Treatment Group — laser in gastric mucosa lesion
  Arms: Laser therapy Treatment Group
Other: Barrier Dust Treatment Group — barrier powder in gastric mucosa lesion
  Arms: Barrier Dust Treatment Group

SUMMARY:
Compare the healing time of lesions in the mucosa of the gastric stoma of children and adolescents using laser therapy versus conventional treatment with protective barrier powder.

DETAILED DESCRIPTION:
Gastrostomy is a procedure indicated for children and adolescents with chronic disease such as intestinal malabsorption, swallowing disorders, neurological diseases, and can progress with peristomal lesions. Thus, it is essential that health professionals know how to take care of ostomies. Today there are several treatments for stoma injuries, however low-level light therapy has been gaining more prominence when we talk about treatment of tissue injury because it is an atraumatic method that, through its analgesic, anti-inflammatory and tissue biomodulation effects, reduces the treatment time of ample spectrum, without causing drug interactions. Therefore, this study seeks to highlight the effect of low-level light therapy on patients. Objective: To compare the healing time of lesions present in the mucosa of the gastric stoma of children and adolescents using laser therapy versus conventional treatment with protective barrier powder. Methodology: randomized, open, comparative clinical trial to assess the healing time of a lesion present in the gastric stoma mucosa using laser therapy or protective barrier powder in a sample of 70 patients aged 0 to 19 years attended by the stoma nurse in the units The work will compare two treatments (two-tailed test), with an alpha error of 5%, and with the power of the 95% test for a means test (Wilcoxon-Mann-Whitney), with an increase of 20% in the sample size, referring to possible losses during the study. The results will be presented as median (variation) or mean ± standard deviation for continuous variables and number (%) for categorical variables. The lesions will be evaluated through an initial measurement and during the treatment days, appearance and number of applications of the laser or protective barrier powder.

ELIGIBILITY:
Inclusion Criteria: children and adolescents from 0 to 19 years old, with lesion in the gastric mucosa regardless of size, hospitalized or undergoing treatment at the Renal Replacement Therapy Unit, who do not present contraindications for phototherapy and who accept to participate in the proposed treatment from the signing of the Age-appropriate consent form and the legal guardian's consent form.

Exclusion Criteria: patients with infection at the application site, with photosensitivity or hypersensitivity caused by laser radiation, with a pacemaker or other electronic implant, patients with malignant lesions or undiagnosed lesion on the area of the stoma to be irradiated, patients and / or legal guardian who does not accept to participate.

Ages: 1 Month to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-08-10 (Actual); Primary Completion 2021-08-10 (Estimated); Study Completion 2023-08-10 (Estimated)

PRIMARY OUTCOMES:
Healing time with laser therapy | 7 days
  Healing time in days of treatment since the first session
Healing time with protective barrier powder | 15 days
  Healing time in days of treatment since the first session

CONTACTS AND LOCATIONS:
Overall Officials: Juliana Ferreira, PhD, Principal Investigator — Instituto da Criança HCFMUSP
Locations (1):
- USaoPauloGH, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No